CLINICAL TRIAL: NCT04815382
Title: Effects of a Dynamic Upper Limb Orthosis in Reducing Tremor and Rigidity on Patients With Parkinson's Disease: a Randomized Clinical Test Study Protocol
Brief Title: Effects of a Dynamic Upper Limb Orthosis in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Burgos (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBU-HUBU: DO
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Tremor, Limb; Rigidity, Muscle
Keywords: Parkinson Disease; Tremor; Rigidity; Upper Limb; Dynamic Orthosis
MeSH Terms: conditions — Parkinson Disease; Tremor; Muscle Rigidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Upper Limb Orthosis group (Experimental): The dynamic upper limb orthosis group will receive a treatment based on the use of a dynamic upper limb orthosis.
  Participants of this group will continue to receive their regular therapy
  Interventions: Other: Dynamic Upper Limb Orthosis
- Control group (No Intervention): The control group will not receive any type of intervention Participants of this group will continue to receive their regular therapy

INTERVENTIONS:
Other: Dynamic Upper Limb Orthosis — The dynamic upper limb orthosis extends from subdeltoid level to 10 mm distal to the metacarpal-phalangeal joints. The orthosis will be tailored to include 20 degrees of wrist extension and to abduct the thumb. They made from nylon and lycra.
  The orthosis will be used throughout the day, being removed when the patient lies down.
  The orthosis will be used during 3 months
  Arms: Dynamic Upper Limb Orthosis group

SUMMARY:
This is a randomized controlled clinical trial aimed at Parkinson's disease patients. Its objective is to evaluate the effects of a dynamic upper limb orthosis to achieve maximum hand functionality, reducing tremor and rigidity

DETAILED DESCRIPTION:
Objective: To assess the effect at 3 and 6 months of the upper limb orthosis, applied for 3 months in the functionality of the affected upper member, manual dexterity, performance of daily living activities and quality of life in Parkinson patients.

Design and setting: A randomized controlled clinical trial of two parallel groups.

Population: 40 patients with tremor and stiffness due to Parkinson´s disease will be included, selected by consecutive sampling at the Neurological Service and Stroke Unit of the Burgos University Hospital (Spain)

. Measurements and intervention: Functionality of the affected upper member, manual dexterity, performance of daily living activities and health-related quality of life will be evaluated. All participants will continue to receive the medical treatment indicated to their health status. The intervention group will receive a treatment based on a dynamic orthosis during 3 months. No additional intervention with the participants of the control group will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to "brain bank" criteria
* Parkinson's disease stage 1 to 3 according to the Hoehn and Yahr scale

Exclusion Criteria:

* Moderate cognitive or language impairment
* Musculoskeletal or dermatological diseases in the upper limb
* Impossibility of follow-up for 6 months
* Difficulty to attend to assessment visits
* Allergy to glove composition

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Rigidity of the upper limb | 3 months
  Measurement by the Movement Disorders. Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Subscale III Score between 0 (best functionality) and 68 (worst functionality)
Tremor of the upper limb | 3 months
  Measurement by the Kinesia One Device This device will provide information on the speed, amplitude and rhythm of the tremor of the upper limb. There are no minimum or maximum values

SECONDARY OUTCOMES:
Manual dexterity of the upper limb | 3 months
  Measurement by the Purdue Pegboard Test Reference values according to age, sex and type of activity
Daily Living Activities | 3 months
  Measurement by the Movement Disorders. Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Subscale II Score between 0 (best functionality) and 52 (worst functionality)
Emotional state and quality of life. | 3 months
  Measurement by the Parkinson's Disease Questionnaire (PDQ-39) The patient points out the frequency of presentation of different situations. It is a quantitative variable; there are no minimum or maximum values; there are no reference values

CONTACTS AND LOCATIONS:
Overall Officials: Raúl Soto-Cámara, PhD, Principal Investigator — University of Burgos; Jeronimo Javier González-Bernal, PhD, Principal Investigator — University of Burgos
Locations (1):
- Universitary of Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No